CLINICAL TRIAL: NCT00501592
Title: An Exploratory Study of INT-747 in Patients With Type 2 Diabetes Mellitus and Presumed Nonalcoholic Fatty Liver Disease
Brief Title: Study of INT-747 in Patients With Diabetes and Presumed NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 747-203
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type II; Fatty Liver
Keywords: Farnesoid X receptor agonist; Metabolic Disorder; Diabetes; NAFLD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatty Liver; Metabolic Diseases; Diabetes Mellitus; Non-alcoholic Fatty Liver Disease | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 25 mg INT-747 (Active Comparator)
  Interventions: Drug: INT-747
- 50 mg INT-747 (Active Comparator)
  Interventions: Drug: INT-747
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INT-747 — 25 mg by mouth once daily, 50 mg by mouth once daily
  Arms: 25 mg INT-747; 50 mg INT-747
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to assess, in patients with Type 2 diabetes mellitus (DM) and presumed nonalcoholic fatty liver disease (NAFLD), the following:

* The safety and tolerability of multiple doses of INT 747;
* The effects of 2 dose levels (25 mg and 50 mg) of INT 747 on insulin resistance and glucose homeostasis;
* Effects of INT-747 on hepatocellular function as measured by assessment of liver enzymes and biochemical markers of hepatic and metabolic function and inflammation, and;
* Trough concentrations of INT-747 and its metabolites, glyco 6-ethyl chenodeoxycholic acid (6-EDCA) and tauro 6-ECDCA.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, placebo-controlled, multiple-dose, parallel-group study. Three (3) cohorts of 12 patients each will receive either placebo, 25 mg INT-747, or 50 mg INT-747 by mouth daily for 6 weeks.

The primary objective of assessing changes in insulin resistance and glucose homeostasis will be attained by performing a euglycemic clamp procedure at baseline (Day 0) and at the end of 6 weeks of treatment (Day 43). Other endpoints will be evaluated by monitoring adverse experiences; vital signs; clinical laboratory values; plasma drug and metabolite concentrations; and general health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, defined by the American Diabetes Association (ADA), as one of the following criteria:
* Symptoms of diabetes plus casual plasma glucose concentration >200 mg/dL (11.1 mmol/L) or
* Fasting plasma glucose >126 mg/dL (7.0 mmol/L) or
* 2-hour post-load glucose >200 mg/dL (11.1 mmol/L) during a 75 g oral glucose tolerance test (GTT).
* Presumed NAFLD, defined by one of the following criteria:
* Alanine aminotransferase (ALT) ≥47 U/L for females and ≥56 U/L for males
* Aspartate aminotransferase (AST) ≥47 U/L for females and ≥60 U/L for males
* Enlarged liver (demonstrated by ultrasound or other imaging technique)
* Diagnostic histological findings shown on prior biopsy (in the last 5 years).

Exclusion Criteria:

* Bilirubin >2 × ULN
* ALT >155 U/L for females and >185 U/L for males.
* AST >155 U/L for females and >200 U/L for males.
* Patients taking any antidiabetic medications, with the exception of metformin and sulfonylureas. If the HbA1c is <11%, patients may be enrolled who have been withdrawn from all other diabetic medications as specified in the protocol, at the discretion of the Principal Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Shapiro, M.D., Study Director — Intercept Pharmaceuticals
Locations (4):
- United States (4):
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - UC San Diego VAMC, San Diego, California
  - Diabetes & Glandular Disease Research Associates, Inc., San Antonio, Texas
  - Virginia Commonwelath University, Richmond, Virginia

REFERENCES:
- [Derived] Mudaliar S, Henry RR, Sanyal AJ, Morrow L, Marschall HU, Kipnes M, Adorini L, Sciacca CI, Clopton P, Castelloe E, Dillon P, Pruzanski M, Shapiro D. Efficacy and safety of the farnesoid X receptor agonist obeticholic acid in patients with type 2 diabetes and nonalcoholic fatty liver disease. Gastroenterology. 2013 Sep;145(3):574-82.e1. doi: 10.1053/j.gastro.2013.05.042. Epub 2013 May 30. PMID 23727264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty four subjects were enrolled in the study at 4 sites. Of the randomized subjects, 20 were randomized to INT-747 25 mg, 21 subjects to INT-747 50 mg, and 23 subjects to placebo. Study enrollment by center ranged from 4 to 31 subjects.
Pre-assignment Details: A protocol amendment allowed for the enrollment of 14 replacement subjects (to enroll up to 56 subjects meeting eligibility requirements). The amendment pre-specified that the original 14 subjects being replaced would not be included in the efficacy analysis since they did not meet the protocol requirements.
Groups:
- 25 mg INT-747; 50 mg INT-747; Placebo: Once daily by mouth
Period: Overall Study
Arm/Group | 25 mg INT-747 | 50 mg INT-747 | Placebo
Started | 20 | 21 | 23
Completed | 20 | 16 | 20
Not Completed | 0 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg INT-747 | 50 mg INT-747 | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 23 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 20 | 59
  >=65 years | 1 | 1 | 3 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 52.7 (8.7) | 50.5 (10.8) | 53.1 (12.1) | 52.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 13 | 31
  Male | 14 | 9 | 10 | 33
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 23 | 64

OUTCOME MEASURES:

1. Primary Outcome: Insulin Resistance and Glucose Homeostasis
Description: The primary objective of assessing changes in insulin resistance and glucose homeostasis will be attained by performing a euglycemic clamp procedure at baseline (Day 0) and at the end of 6 weeks of treatment (Day 43).
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | 25 mg INT-747 | 50 mg INT-747 | Placebo
Number analyzed (Participants) | 20 | 21 | 23
mg/kg/min
  Low Dose Insulin | .69 (1.12) | .24 (1.62) | -0.51 (1.88)
  High Dose Insulin | .73 (1.53) | .42 (1.42) | -0.61 (1.88)
Statistical Analysis 1: Comparison: 25 mg INT-747 vs Placebo; The primary endpoints are calculated as the change (post minus pre treatment) during low dose and high dose insulin infusion periods. These are compared between placebo and INT-747 25 mg using t-tests for independent samples. These tests will be made without correction for multiple comparisons using 0.05 as the alpha criterion for significance. Results will be described with the corresponding means and standard deviations; Test type: Superiority or Other; p = 0.040, t-test, 2 sided
Statistical Analysis 2: Comparison: 50 mg INT-747 vs Placebo; The primary endpoints are calculated as the change (post minus pre treatment) during low dose and high dose insulin infusion periods. These are compared between placebo and INT-747 50 mg using t-tests for independent samples. These tests will be made without correction for multiple comparisons using 0.05 as the alpha criterion for significance. Results will be described with the corresponding means and standard deviations; Test type: Superiority or Other; p = 0.28, t-test, 2 sided

2. Secondary Outcome: Hepatocellular Function
Description: Hepatocellular function as measured by assessment of liver enzymes and biochemical markers of hepatic and metabolic function
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 25 mg INT-747 | 50 mg INT-747 | Placebo
Number analyzed (Participants) | 20 | 21 | 23
U/L
  ALT | -9 (14) | 9 (47) | 11 (48)
  AST | -3 (7) | 4 (24) | 4 (46)
  GGT | -39 (77) | -23 (56) | 5 (27)
Statistical Analysis 1: Comparison: 25 mg INT-747 vs Placebo; Test type: Superiority or Other; p = 0.0031, t-test, 2 sided
Statistical Analysis 2: Comparison: 50 mg INT-747 vs Placebo; Test type: Superiority or Other; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: 25 mg INT-747 vs Placebo; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: 50 mg INT-747 vs Placebo; Test type: Superiority or Other; p = 0.0005, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: One year, 7 monhts
Arm/Group | 25 mg INT-747 | 50 mg INT-747 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 6/20 | 15/21 | 13/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg INT-747 (N=20) | 50 mg INT-747 (N=21) | Placebo (N=23)
Vessel Puncture Site Pain (General disorders) | 1 (1) | 4 (6) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 3 (5) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed publications based on this study shall be approved by the Sponsor prior to submission for publication. Such approval will not be unreasonably witheld. Publications will reflect the contributions made by the Investigators, Sponsor personnel and other groups involved in the study.